CLINICAL TRIAL: NCT04559009
Title: COVID-19 Amyotrophic Lateral Sclerosis (ALS) Registry
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00082131; AH-NSI-COVID19-ALS (Other: Atrium)
Record Dates: First submitted 2020-09-21; First posted 2020-09-22 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Covid19; Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — COVID-19; Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a relentlessly progressive and fatal neurodegenerative disease characterized by progressive weakness involving limb, bulbar, and respiratory muscles.There is currently no information suggesting how COVID-19 affects patients diagnosed with amyotrophic lateral sclerosis (ALS). This is especially important as respiratory compromise is common in ALS patients and can complicate the clinical course as COVID-19 could lead to respiratory failure and need for intubation. We intend that this registry will guide our understanding of how COVID-19 affects patients with ALS.

DETAILED DESCRIPTION:
The purpose of this registry is to assess the incidence and prevalence of COVID-19 in ALS patients, the effect of COVID-19 on ALS disease trajectory, and the impact, if any, of edaravone, riluzole and other concomitant medication used in ALS like Albuterol and dextromethorphan/quinidine (Nuedexta) on these parameters. COVID-19 incidence and prevalence in the ALS population will be assessed through outcomes reporting ranging from recovered infections to patient death reported in a patient facing registry.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ALS and
* A confirmed COVID-19 infection determined by:

  1. positive SARS-CoV-2 viral RNA PCR test and/or
  2. positive serology antibody testing for SARS-CoV-2

Exclusion Criteria:

* No ALS diagnosis
* No confirmed COVID-19 infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our study population consists of qualifying cases of patients with ALS who have had a laboratory confirmed COVID-19 infection.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
COVID-19 incidence and prevalence in the ALS population | Data will be collected through study completion, an average of 3 years
  Assessed through outcomes reporting ranging from recovered infections to patient death reported in a patient facing registry.

CONTACTS AND LOCATIONS:
Overall Officials: Urvi Desai, MD, Principal Investigator — Neurologist/ MDA Director
Locations (1):
- Neurosciences Institute, Neurology - Charlotte, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No